CLINICAL TRIAL: NCT04712890
Title: A Multi-center, Non-interventional, Prospective Cohort Study for Determination of Prevalence and Features of HRRm mCRPC (ADAM)
Brief Title: Determination of Prevalence and Features of HRRm mCRPC (ADAM)
Acronym: ADAM
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D133HR00008
Record Dates: First submitted 2021-01-08; First posted 2021-01-15 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: HRRm mCRPC
Keywords: HRRm mCRPC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Study design:

This study is local, multi-center, prospective, cohort study to collect real world data related mCRPC patients, prevalence of HRRm and to assess possible influence of HRRm on treatment outcomes. No additional procedures besides those already used in the routine clinical practice will be applied to the patients. Treatment assignment will be done according to the current practice.

Data Source(s):

For testing archival samples (formalin fixed and paraffin embedded [FFPE]) from primary tumor will be used . 15 HRR genes (BRCA1, BRCA2, ATM, BRIP1, BARD1, CDK12, CHEK1, CHEK2, FANCL, PALB2, PPP2R2A, RAD51B, RAD51C, RAD51D and RAD54L) will be analyzed using NGS in dedicated central laboratory facilities. Choice of laboratory for each center will be made based on logistical proximity. Each NGS laboratory will have to determine and report clinical significance of alterations found using database search or other predictors to classify variants as deleterious or suspected deleterious. VUS have to be reported separately. Benign variants will be not reported in this study.

All clinical and demographic data for patients with finished therapy will be collected in prospective or retrospective (where applicable) manner during the study visits. The second visit will take place when the disease progression or death is occurs or in a year after the first visit whichever happens first. Data will be entered in the eCRF. The site investigator will be responsible for ensuring that all required data is collected and entered into the eCRF with the involvement of clinical research organization.

It is estimated that approximately 300 patients will be enrolled in the first stage. After interim analysis total number of the patients can be increased, depending on the number of NGS failures. It is estimated that approximately 30 sites in total will be participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male 18 years age or older
* Provision of written informed consent
* Histologically confirmed diagnosis of prostate cancer
* Documented evidence of metastatic castration resistant prostate cancer (mCRPC)
* Patients who are on the first line therapy or already received one line of therapy due to mCRPC previously
* Availability of archival FFPE tissue from primary prostate tumor
* Availability of medical history (e.g. out-patient medical records or disease histories for hospitalized patients)

Exclusion Criteria:

• Patients participating in clinical studies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of mCRPC patients with available medical history and FFPE specimen of archival tissue from primary prostate tumor and who received at least one line of therapy for mCRPC or is currently receiving this therapy. It is estimated that 300 patients will be enrolled (this sample can be further increased after the interim analysis based on the actual number of NGS failures). It is estimated that approximately 30 sites in total will be participating in the study. There will be 2 cohorts of patients: HRRm and HRRwt to reveal possible differences in treatment pattern, demographic and clinical characteristics and outcomes in mCRPC patients with and without HRRm.
Sampling Method: Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Differences in demographics between patients with HRRm and HRRwt mCRPC | Up to 1 year
Differences in treatment patterns between patients with HRRm and HRRwt mCRPC | Up to 1 year
Differences in clinical characteristics between patients with HRRm and HRRwt mCRPC | Up to 1 year
Progression-free survival (PFS) rate (time to documentation of objective tumor progression/relapse) stratified by tissue HRR-related gene mutation status and by treatment pattern | Up to 1 year

CONTACTS AND LOCATIONS:
Locations (14):
- Russia (14):
  - Research Site, Barnaul, Altayskiy Kray
  - Research Site, Ufa, Bashkortostan Republic
  - Research Site, Chelyabinsk, Chelyabinsk Oblast
  - Research Site, Krasnoyarsk, Krasnoyarsk Krai
  - Research Site, Saint Petersburg, Leningradskaya Oblast'
  - Research Site, Nizhny Novgorod, Nizhniy Novgorod Region
  - Research Site, Omsk, Omsk Oblast
  - Research Site, Vladivostok, Primorskiy (Maritime) Kray
  - Research Site, Yuzhno-Sakhalinsk, Sakhalin Oblast
  - Research Site, Yekaterinburg, Sverdlovsk Oblast
  - Research Site, Tyumen, Tyumen Oblast
  - Research Site, Yaroslavl, Yaroslavl Oblast
  - Research Site, Moscow
  - Research Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: Redacted CSR synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D133HR00008&attachmentIdentifier=b6324e74-e298-4ba5-9d41-5c03357da902&fileName=D133HR00008_Study_report_Synopsis_Redacted.pdf&versionIdentifier=